CLINICAL TRIAL: NCT06242782
Title: Vertical Ridge Augmentation Strategies: An Adaptive Randomised Controlled Clinical Trial
Brief Title: Vertical Ridge Augmentation Strategies
Acronym: VARGAS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS ID 297914; IRAS ID 297914 (Other: Integrated Research Application System); EDGE ID 144889 (Other: UCLH and UCL's study and trial management system)
Record Dates: First submitted 2024-01-05; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Alveolar Bone Resorption; Alveolar Ridge Trauma; Alveolar Bone Loss; Complication of Surgical Procedure
Keywords: Vertical Ridge Augmentation; Vertical Bone Augmentation; Alveolar Bone Grafting
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Positive Control (Active Comparator): VRA using Ti-Reinforced d-PTFE membrane
  Interventions: Procedure: VRA + d-PTFE membrane
- Test 1 (Experimental): VRA using Ti-Reinforced e-PTFE membrane
  Interventions: Procedure: VRA + e-PTFE membrane
- Test 2 (Experimental): VRA using 3D printed Titanium mesh
  Interventions: Procedure: VRA + customised Ti-mesh
- Test 3 (Experimental): VRA using Reinforced PTFE mesh
  Interventions: Procedure: VRA + RPM

INTERVENTIONS:
Procedure: VRA + d-PTFE membrane — VRA using a 50/50 particulate bone mix (xenograft+ autograft) + Ti-Reinforced d-PTFE membrane
  Arms: Positive Control
Procedure: VRA + e-PTFE membrane — VRA using a 50/50 particulate bone mix (xenograft+ autograft) + Ti-Reinforced e-PTFE membrane
  Arms: Test 1
Procedure: VRA + customised Ti-mesh — VRA using a 50/50 particulate bone mix (xenograft+ autograft) + 3D printed Titanium mesh
  Arms: Test 2
Procedure: VRA + RPM — VRA using a 50/50 particulate bone mix (xenograft+ autograft) + Reinforced PTFE mesh
  Arms: Test 3

SUMMARY:
Guided Bone Regeneration (GBR) is an invaluable and beneficial surgical technique adopted when there is the need to augment an alveolar atrophy. Strong clinical and histologic evidence exists on the effectiveness and predictability of GBR in bone augmentation of ridge deficiencies. On the other hand, it is well known that GBR remains a challenge as in the most extreme cases, it is considered a highly technique-sensitive surgical procedure.

Whilst there are numerous reviews which report the average incidence of complications in GBR, there is still insufficient evidence and manuscripts reporting a direct correlation between a specific biomaterial (membrane or scaffold) and observed complications. Only one recent systematic review and meta-analysis focused on wound healing complications following GBR for ridge augmentation procedures. Authors explored the complication rate based on the membrane type and on the timing of the first sign of soft tissue complications following bone augmentation procedures. They reported a complication rate of 17% of the overall soft tissue complications, including membrane exposure, soft tissue dehiscence, and acute infection (abscess). This estimate is consistent with that reported (12%) in a more recent systematic appraisal of the evidence on all types of complications in GBR (3). However, when horizontal augmentation procedures were reviewed, a higher rate (21%) of complications was reported within the first 18 months of a GBR procedure. This estimate was inclusive of all possible biologic complications following GBR whilst the rate of membrane exposure was of 23%.

Vertical bone augmentation represents one of the most challenging bone regenerative procedures in surgical dentistry. This is because of the inherent difficulties of the surgical procedure and the high risk of complications. The primary aim of this procedure is to recreate alveolar bone in a vertical direction (without the support of any pre-existing walls) and enable recreation of a more favourable anatomy for the restoration of the edentulous site.

Evidence on a variety of treatment options has been produced over the last 15 years including distraction osteogenesis, onlay bone grafting, and vertical ridge augmentation (VRA). Systematic reviews evaluating the efficacy of different surgical procedures for VRA either in a staged or a simultaneous fashion, reported a range of vertical bone gain of 2-8 mm. This gain was gradually lost (1.27 to 2.0mm) between 1 to 7 years post-surgery and a wide range of complications (0- 45.5%) has been reported.

The aim of this study is to assess and compare incidence of complications and percentage of vertical bone gain when using four different barrier membranes in combination with 50/50 autogenous and xenogenous bone material in VRA procedures. Secondary aims will be to evaluate and compare early and late soft tissue wound healing, gingival microvasculature and structure, patient reported outcomes and the prevalence of need for further bone augmentation and need for soft tissue grafting. Additionally, this study will also aim to assess and compare histomorphometry and histochemistry analyses of core biopsies obtained before implant placement between the four different barrier membranes.

DETAILED DESCRIPTION:
This is a single centre non-inferiority adaptive randomised controlled clinical trial. The primary aim of this study will be:

To assess the clinical composite outcome (incidence of complications and percentage of vertical bone gain) of vertical alveolar bone grafting procedures in patients with vertical ridge deficiencies prior to dental implant placement, using a mix of autogenous and xenogenic particulate bone materials in combination with four different barrier membranes (Titanium (Ti)-Reinforced d-Polytetrafluoroethylene (PTFE) membrane [control group], Ti-Reinforced e-PTFE Membrane, 3D printed Ti-mesh and Reinforced PTFE Mesh (RPM)).

Secondary aims are:

* To assess and compare soft tissue wound healing and vascularization using Laser Doppler Flowmetry (LDF) between tests and control.
* To assess and compare gingival microvasculature and structure in vivo using Optical Coherence Tomography (OCT) between tests and control.
* To compare prevalence of the need for further bone grafting at the time of implant placement between tests and control.
* To compare prevalence of the need of soft tissue grafting at second stage surgery between tests and controls.
* To assess and compare patient reported outcomes using the EuroQol five-dimension (EQ-5D-5L) scale and the short-form Oral Health Impact Profile (OHIP-14) between tests and control.
* To assess and compare histomorphometry and histochemistry analyses of core biopsies obtained from a sample of 5 participants from each group before implant placement between tests and control.

Patients in need of vertical ridge augmentation prior to dental implant placement will be recruited to take part in this study and will be randomised into one of the following groups receiving different interventions:

1. VRA using a 50/50 particulate bone mix (xenograft+ autograft) + Ti-Reinforced d- PTFE membrane (Positive Control)
2. VRA using a 50/50 particulate bone mix (xenograft+ autograft) + Ti-Reinforced e-PTFE membrane (Test 1).
3. VRA using a 50/50 particulate bone mix (xenograft+ autograft) + 3D printed Titanium mesh (Test 2).
4. VRA using a 50/50 particulate bone mix (xenograft+ autograft) + Reinforced PTFE mesh (Test 3)

One-hundreds and forty-eight (148) participants meeting inclusion/exclusion criteria and who consent to this study will undergo a baseline visit assessment (visit 2) in which they will have a comprehensive oral assessment, radiographic assessment of alveolar defect using Cone Beam CT and supportive periodontal therapy. After randomisation to either Tests (1-3) or Control Groups, each group will undergo a VRA procedure as randomised (visit 3). All patients will be re-examined at 1, 3, 7, 15, 30, 60 and 120 days (visits 4-10, respectively) after the surgical augmentation. At each assessment, clinical examination, soft tissue imaging measures and saliva collections will be performed. Additionally, supportive periodontal therapy will be provided to all participants at the 120 days post augmentations visit. All participants will then undergo dental Implants placement after 180 days (visit 11). Participants will then be followed at 7, 15, 30,90, 120, 180 and 365 days (visits 12-18) after dental implant placement. The 90 days post implantation visit will include supportive periodontal therapy while the 120 days visit will involve the placement of dental implant prosthetic components for all participants.

Statistical methodology and analysis:

Primary and secondary outcomes analysis:

Continuous data are displayed as mean and standard deviation whilst categorical variables will be reported as percentages and prevalence. All participants randomized to test or control will be included in final analyses. Analysis will be performed using last observation carrying forward and as intent to treat population. Secondarily, per protocol analysis will also be performed. Data will be entered in an electronic spreadsheet and checked/proofed for any errors. All data will be loaded in the appropriate software for analysis. The primary outcome assessment will be assessed by analysis of co-variance model. Age, gender, body mass index and ethnicity will be included as principal covariates. Pair-wise comparison and between groups differences will be calculated using Tukey corrections.

All secondary endpoints will be analysed in a similar fashion. Significance will be set to be at p ≤ 0.05. Adverse events analysis will also be performed between study groups at study visits. Serial changes in imaging variables will be analysed with analysis of variance for repeated measures using a conservative F-test (Greenhouse-Geisser correction). If a treatment by time interaction will be found, pair-wise comparisons will be performed (Bonferroni-Holm adjustment).

Sensitivity and other planned analyses:

In this trial, investigators will perform some types of the sensitivity analysis, including non-statistical and statistical analyses. The sensitivity analysis that investigators will be including are impact of non-compliance/protocol deviation, impact of missing data, impact of competing risk in analysis of composites outcomes, impact of baseline imbalance, and finally, related to statistical analysis is impact of different assumptions underlying statistical model. The option plan for the condition related to non-compliance/protocol deviation are intention-to-treat (ITT) analysis; as per protocol analysis; and as-treated analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Partially edentulous with a ridge that shows at least 3mm vertical bone deficiency;
2. Females of childbearing potential and males agree to use an effective method of contraception from the time consent is signed until treatment discontinuation.
3. Females of childbearing potential have a negative pregnancy test within 7 days prior to being registered. Participants are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Comorbidities (or regular use of medications)
2. History of bone augmentation or implant placement at the area of interest
3. Females who are pregnant, planning pregnancy or breastfeeding
4. Regular use of analgesic or antibiotics within 1 month before entering the study
5. Disclosed smoking (including electronic cigarettes) or drinking over 14 alcoholic units per week
6. Active oral diseases or poor oral hygiene (defined by full mouth dental plaque scores greater than 25%)
7. Suspected or documented titanium allergy or intolerance
8. Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within last 3 months of study enrolment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | Baseline visit (day 0) and follow up visits (at days 1, 4(±1), 7(±1), 15(±1), 30(±3), 60(±7) and 120(±7) post surgical VRA and at days 7(±1), 15(±1), 30(±7), 90(±7), 120(±7), 180 (±14) and 365 (±14) post dental implant placement
  Measured by clinical observation/examination at each follow up visit following VRA surgery.
Percentage of vertical bone gain | At baseline (before surgical VRA) and at time of dental implant(s) placement (not earlier than 180 days post surgical VRA)
  Measured on cone beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Soft tissue vascularization and wound healing | Baseline visit (day 0) and follow up visits (at days 1, 4(±1), 7(±1), 15(±1), 30(±3), 60(±7) and 120(±7) post surgical VRA and at days 7(±1), 15(±1), 30(±7), 90(±7), 120(±7), 180 (±14) and 365 (±14) post dental implant placement
  Measured by Laser Doppler Flowmetry (LDF).
Gingival microvasculature and structure in vivo | Baseline visit (day 0) and follow up visits (at days 1, 4(±1), 7(±1), 15(±1), 30(±3), 60(±7) and 120(±7) post surgical VRA and at days 7(±1), 15(±1), 30(±7), 90(±7), 120(±7), 180 (±14) and 365 (±14) post dental implant placement
  Measured by Optical Coherence Tomography (OCT)
Need for additional bone grafting | At time of dental implant(s) placement (not earlier than 180 days post surgical VRA)
Need of soft tissue grafting | At time of dental implant(s) placement (not earlier than 180 days post surgical VRA)
Patient reported outcome measures | Baseline visit (day 0) and follow up visits (at days 1, 4(±1), 7(±1), 15(±1), 30(±3), 60(±7) and 120(±7) post surgical VRA and at days 7(±1), 15(±1), 30(±7), 90(±7), 120(±7), 180 (±14) and 365 (±14) post dental implant placement
  Using the 5-level EQ-5D (EQ-5D-5L). The EQ-5D-5L scores can range from <0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Patient reported outcome measures | Baseline visit (day 0) and follow up visits (at days 1, 4(±1), 7(±1), 15(±1), 30(±3), 60(±7) and 120(±7) post surgical VRA and at days 7(±1), 15(±1), 30(±7), 90(±7), 120(±7), 180 (±14) and 365 (±14) post dental implant placement
  Using the short-form Oral Health Impact Profile (OHIP-14). The OHIP-14 scores can range from 0 to 56. Higher scores indicate worse and lower scores indicate better Oral Health Related Quality of Life.
Histomorphometry analysis | At time of dental implant(s) placement (not earlier than 180 days post surgical VRA)
  Using core biopsies obtained from a sample of 5 participants from each group
Histochemistry analysis | At time of dental implant(s) placement (not earlier than 180 days post surgical VRA)
  Using core biopsies obtained from a sample of 5 participants from each group

CONTACTS AND LOCATIONS:
Overall Officials: Francesco D'Aiuto, Principal Investigator — University College, London

IPD SHARING:
Plan to Share IPD: No
Could be available upon reasonable request

REFERENCES:
- [Result] Alotaibi FF, Rocchietta I, Buti J, D'Aiuto F. Comparative evidence of different surgical techniques for the management of vertical alveolar ridge defects in terms of complications and efficacy: A systematic review and network meta-analysis. J Clin Periodontol. 2023 Nov;50(11):1487-1519. doi: 10.1111/jcpe.13850. Epub 2023 Jul 26. PMID 37495541
- [Result] Rocchietta I, Simion M, Hoffmann M, Trisciuoglio D, Benigni M, Dahlin C. Vertical Bone Augmentation with an Autogenous Block or Particles in Combination with Guided Bone Regeneration: A Clinical and Histological Preliminary Study in Humans. Clin Implant Dent Relat Res. 2016 Feb;18(1):19-29. doi: 10.1111/cid.12267. Epub 2015 Jan 27. PMID 25622713